CLINICAL TRIAL: NCT01208974
Title: A Phase I Trial Assessing the Safety and Feasibility of Prophylactic Nipple-Areola Complex (NAC) Irradiation After Nipple-Sparing Mastectomy and Immediate Reconstruction in Patients With In-Situ or Invasive Breast Cancer
Brief Title: Nipple-Areola Complex (NAC) Irradiation After Nipple-Sparing Mastectomy and Reconstruction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Cristiane Takita, Professor of Clinical, University of Miami
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20090299; SCCC-2009004 (Other: University of Miami Sylvester Comprehensive Cancer Center)
Record Dates: First submitted 2010-09-22; First posted 2010-09-24 (Estimated); Results first posted 2022-01-18 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Ductal Carcinoma
Keywords: Breast Cancer; Nipple Area Complex; Mastectomy; Radiation Therapy; Nipple-Sparing; Breast Reconstruction
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Ductal | interventions — Mastectomy, Subcutaneous; Mammaplasty; Sentinel Lymph Node Biopsy

STUDY DESIGN:
Intervention Model Description: Phase 1 dose-escalation/de-escalation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Phase 1 MTD NAC RT (Experimental): Participants will undergo a Nipple-Areolar Complex (NAC)-sparing mastectomy with immediate reconstruction and axillary surgery, if indicated, on Week 1. Anytime between Weeks 5-8, participants will undergo a dose-escalation/de-escalation of prophylactic NAC radiation treatment (RT) twice daily (minimum of 4 hours apart) for 5 days. Dose escalation/de-escalation design are as follows:
  * Dose Level I - 10 fractions of 2.0 Gy for a total of 20 Gy
  * Dose Level II - 10 fractions of 2.5 Gy for a total of 25 Gy
  * Dose Level III - 10 fractions of 3.0 Gy for a total of 30 Gy
  * Dose Level IV - 10 fractions of 3.5 Gy for a total of 35 Gy
  Participants will be treated between cohorts of 2-6 patients per dose level starting at dose level II. Dose escalation stops when 2 out of 2-6 participants encounter Dose Limiting Toxicities (DLT).
  Standard of care chemotherapy, at treating physician's discretion, can be initiated 2 weeks after RT.
  Interventions: Procedure: Nipple-Sparing Mastectomy; Procedure: Breast Reconstruction; Procedure: Axillary Surgery; Radiation: Prophylactic Nipple-Areolar Complex RT

INTERVENTIONS:
Procedure: Nipple-Sparing Mastectomy — Subcutaneous Mastectomy (SCM) to be performed, preserving the nipple and areola complex, after a frozen section of the tissue underneath the nipple-areola complex is sampled and found to be negative for tumor. Performed during Week 1.
  Other Names: NAC-sparing mastectomy; Nipple and areola complex-sparing mastectomy
Procedure: Breast Reconstruction — Immediate reconstruction of the breast will be performed (after Nipple-Sparing Mastectomy) by the plastic surgeon, type depend on surgeon's discretion and patient's desire. Performed during Week 1.
Procedure: Axillary Surgery — Axillary Dissection or Sentinel Node Biopsy (SNB) will be performed at surgeon's discretion.
  Other Names: Axillary Dissection; Sentinel Node Biopsy
Radiation: Prophylactic Nipple-Areolar Complex RT — Prophylactic Nipple-Areolar Complex Radiation Therapy per protocol. Administered between weeks 5 to 8.
  Other Names: Prophylactic NAC Radiation Therapy

SUMMARY:
The purpose of this research study is to see if a participant's nipple and areola can be safely preserved by adding radiation to these areas after a nipple-sparing mastectomy and immediate breast reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed in-situ or invasive breast carcinoma.
* Tis, T1, T2 invasive or non-invasive carcinoma of the breast; lesion less than 4 cm.
* Unifocal, multifocal or multicentric breast cancers that can be removed by nipple sparing mastectomy with negative surgical margins.
* No extensive intraductal component or patient with distant metastases.
* Patients must be > 18 years of age.
* No concomitant or history of nipple discharge or skin involvement.
* No prior history of malignancy (less than 5 years prior to study entry), except non-melanomatous skin cancer.
* No prior history of radiation to the chest.
* No collagenous disease (systemic lupus erythematosis, scleroderma, dermatomyositis)No previous non-hormonal therapy including radiation or chemotherapy for current breast cancer.
* No patients with Paget's disease of the nipple.
* No patients with co-existing medical conditions with life expectancy < 2 years.
* No pregnant or lactating women.
* Eastern Cooperative Oncology Group (ECOG) 0 - 2.
* Signed study-specific informed consent form prior to the study entry.

Exclusion Criteria:

* Retroareolar breast cancer lesions within one cm, depth from the skin surface.
* Concomitant or history of nipple discharge or skin involvement.
* Patient with distant metastases.
* Patient with extensive intraductal carcinoma.
* Any previously irradiated ipsilateral breast cancer.
* Patients with Paget's disease of the nipple.
* Patients with collagenous diseases, as systemic lupus erythematosis, scleroderma or dermatomyositis.
* Other malignancy, except nonmelanomatous skin cancer, less than 5 years prior to participation in this study.
* Patients who are pregnant or lactating due to potential exposure of the fetus to RT and unknown effects of RT to lactating females.
* Positive surgical margins following nipple sparing mastectomy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-03-16 (Actual); Primary Completion 2018-02-13 (Actual); Study Completion 2026-05-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Cristiane Takita, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants undergo NAC-Sparing Mastectomy, and then receive prophylactic radiation therapy according to a dose-escalation/de-escalation design, the first cohort of 2 to 6 patients starting at dose level II (10 Fractions of 2.5 Gy). If 2 or more participants experience dose-limiting toxicities at the starting dose level (dose level II), then de-escalation occurs to dose level I (10 Fractions of 2.0 Gy) for the next cohort of 2 to 6 participants. No participants were assigned to dose level I.
Groups:
- NAC-Sparing Mastectomy: Participants who completed Nipple-Areolar Complex (NAC)-sparing mastectomy with immediate reconstruction and axillary surgery, and intra-/post-operative period from weeks 1 to 4. All participants complete this surgery and post-mastectomy period before being assigned to a dosing arm for prophylactic radiation therapy.
- Prophylactic NAC RT - Dose Level II - 10 Fractions of 2.5 Gy (Starting Dose): The first 6 participants that had received the starting dose of NAC Prophylactic Radiation Therapy (RT) at Dose Level II - 10 fractions of 2.5 Gy for a total of 25 Gy after completing NAC-Sparing mastectomy.
- Prophylactic NAC RT - Dose Level III - 10 Fractions of 3.0 Gy: The second group of 6 participants that had received Prophylactic NAC Radiation Therapy (RT) at Dose Level III - 10 fractions of 3.0 Gy for a total of 30 Gy after completing NAC-Sparing mastectomy, and after the first 6 participants reported 0 dose-limiting toxicities (DLTs) at Dose Level II.
- Prophylactic NAC RT - Dose Level IV - 10 Fractions of 3.5 Gy: The third group of 6 participants that had received Prophylactic NAC Radiation Therapy (RT) at Dose Level IV - 10 fractions of 3.5 Gy for a total of 35 Gy after completing NAC-Sparing mastectomy, and after the second 6 participants reported 0 dose-limiting toxicities (DLTs) at Dose Level III.
Period: NAC-Sparing Mastectomy
Arm/Group | NAC-Sparing Mastectomy | Prophylactic NAC RT - Dose Level II - 10 Fractions of 2.5 Gy (Starting Dose) | Prophylactic NAC RT - Dose Level III - 10 Fractions of 3.0 Gy | Prophylactic NAC RT - Dose Level IV - 10 Fractions of 3.5 Gy
Started | 21 | 0 | 0 | 0
Completed | 21 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Post-Mastectomy Period (Weeks 1 to 4)
Arm/Group | NAC-Sparing Mastectomy | Prophylactic NAC RT - Dose Level II - 10 Fractions of 2.5 Gy (Starting Dose) | Prophylactic NAC RT - Dose Level III - 10 Fractions of 3.0 Gy | Prophylactic NAC RT - Dose Level IV - 10 Fractions of 3.5 Gy
Started | 21 | 0 | 0 | 0
Completed | 18 | 0 | 0 | 0
Not Completed | 3 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Period: Prophylactic NAC RT (Weeks 5 to 8)
Arm/Group | NAC-Sparing Mastectomy | Prophylactic NAC RT - Dose Level II - 10 Fractions of 2.5 Gy (Starting Dose) | Prophylactic NAC RT - Dose Level III - 10 Fractions of 3.0 Gy | Prophylactic NAC RT - Dose Level IV - 10 Fractions of 3.5 Gy
Started | 0 | 6 | 6 | 6
Cohort 1: Starting Dose | 0 | 6 | 0 | 0
Cohort 2: 1st Dose Escalation | 0 | 0 | 6 | 0
Cohort 3: 2nd Dose Escalation | 0 | 0 | 0 | 6
Completed | 0 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Phase 1 MTD NAC RT
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Prophylactic NAC Irradiation.
Description: The recommended Phase II dose will be reported as the MTD at which only 0 or 1 out of 6 participants experiences dose limiting toxicity (DLT). DLT will be reported as any of the following: Grade 4 skin rash or pain, NAC necrosis, any toxicity requiring interruption of NAC irradiation greater than 2 weeks or any grade 4 or 5 treatment related toxicity. Toxicity will be evaluated by treating physician using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 3.0.
Time Frame: Up to 13 weeks
Population: A total of 18 participants at dose-escalating study design (6 participants at each dose level - Levels II, III and IV) who received prophylactic NAC RT after nipple-sparing mastectomy were evaluated to assess the MTD/Recommended Phase II dose.
Measure: Number; unit: Gy (grays)
Groups:
- Prophylactic NAC RT After Nipple-Sparing Mastectomy: Participants who received NAC RT after nipple-sparing mastectomy at the following dose levels:
  * Dose Level II: 6 participants receiving 10 fractions at 2.5 grays (gy) for total of 25 Gy.
  * Dose Level III: 6 participants receiving 10 fractions at 3.0 grays (gy) for total of 30 Gy.
  * Dose Level IV: 6 participants receiving 10 fractions at 3.5 grays (gy) for total of 35 Gy.
Arm/Group | Prophylactic NAC RT After Nipple-Sparing Mastectomy
Number analyzed (Participants) | 18
Gy (grays) | 35

2. Secondary Outcome: Cosmetic Outcome
Description: Cosmetic Outcome will be reported as the number of participants in each of the 4 cosmetic outcome category ordinal scale. The 4 cosmetic outcome category scales are excellent, good, fair and poor. Both physician and patient's evaluation will be reported.
Time Frame: 12 months
Reporting Status: Not Posted, anticipated posting 2027-05

3. Secondary Outcome: Disease-Free Survival Rate in Study Participants
Description: Disease-free survival rate in study participants will be assessed. Disease-free survival is defined from the date of surgery until the date of documented recurrence (local or distant) or breast cancer-related death, whichever occurs first. Patients who die without documentation of recurrence will be considered to have had disease recurrence at the time of death, unless there is documented evidence that no recurrence occurred before death.
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2027-05

4. Secondary Outcome: Overall Survival Rate in Study Participants
Description: Overall Survival rate in study participants will be assessed. Overall survival is the defined from the date of surgery until the date of death due to any cause. In the absence of death, follow-up time will be censored by the date of last contact..
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2027-05

5. Secondary Outcome: Recurrence Rate in Study Participants
Description: Rate of disease recurrence in study participants. The definition of local recurrence is histologic evidence of recurrent carcinoma, either invasive or non-invasive in the nipple-areola complex in the ipsilateral breast. Clinical evidence of carcinoma by physical exam and/or mammograms/MRI will not be evidence of local recurrence until biopsy proof.
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2027-05

ADVERSE EVENTS:
Time Frame: Up to 8 months
Groups:
- NAC-Sparing Mastectomy: Participants who completed Nipple-Areolar Complex (NAC)-sparing mastectomy with immediate reconstruction and axillary surgery, and intra-/post-operative period from weeks 1 to 4.
- Prophylactic NAC RT - Dose Level II - 10 Fractions of 2.5 Gy: The first 6 participants that had received the starting dose of NAC Prophylactic Radiation Therapy (RT) at Dose Level II - 10 fractions of 2.5 Gy for a total of 25 Gy after completing NAC-Sparing mastectomy.
Arm/Group | NAC-Sparing Mastectomy | Prophylactic NAC RT - Dose Level II - 10 Fractions of 2.5 Gy | Prophylactic NAC RT - Dose Level III - 10 Fractions of 3.0 Gy | Prophylactic NAC RT - Dose Level IV - 10 Fractions of 3.5 Gy
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/21 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 12/21 | 6/6 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NAC-Sparing Mastectomy (N=21) | Prophylactic NAC RT - Dose Level II - 10 Fractions of 2.5 Gy (N=6) | Prophylactic NAC RT - Dose Level III - 10 Fractions of 3.0 Gy (N=6) | Prophylactic NAC RT - Dose Level IV - 10 Fractions of 3.5 Gy (N=6)
Surgery/Intra-Operative Injury (Surgical and medical procedures) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pain - Other (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NAC-Sparing Mastectomy (N=21) | Prophylactic NAC RT - Dose Level II - 10 Fractions of 2.5 Gy (N=6) | Prophylactic NAC RT - Dose Level III - 10 Fractions of 3.0 Gy (N=6) | Prophylactic NAC RT - Dose Level IV - 10 Fractions of 3.5 Gy (N=6)
Anorexia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back Pain (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Breast Pain (General disorders) | 9 (10) | 1 (1) | 0 (0) | 1 (1)
Chest Wall Pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Depression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis: Radiation (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 4 (4) | 6 (8)
Small area of scab on the left nipple (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin sloughing (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nipple congestion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nipple eschar (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Occasional tightness in the axillary redion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Crusting on incisions (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Burning sensation along the incisions (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Right nipple with slight bulla (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin necrosis (on the side of right prophylactic reconstructed breast) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left breast skin necrosis cancer side (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema: trunk/genital (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5) | 5 (5) | 3 (3)
Insomnia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Breast nipple/areolar deformity (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Occasional pain in the axillary region (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain of skin (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Infection with unknown ANC
Seroma (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Infection with normal ANC or Grade 1 or 2 neutrophils
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vasculitis (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bruising (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — Bruising (in absence of Grade 3 or 4 thrombocytopenia)
Hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT01208974/Prot_SAP_000.pdf